CLINICAL TRIAL: NCT01474382
Title: A Phase 4, Multicenter, Randomized, Double-Blinded, Controlled Study of OraVerse® for Safety and Efficacy in Pediatric Dental Patients Undergoing Mandibular and Maxillary Procedures
Brief Title: Study of OraVerse® for Safety and Efficacy in Pediatric Dental Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novocol Pharmaceutical of Canada, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PHE-11-001
Record Dates: First submitted 2011-11-11; First posted 2011-11-18 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Dental Anesthesia; Anesthesia, Local; Anesthesia, Reversal
Keywords: OraVerse; Safety; Efficacy; Pediatric; Reversal of dental anesthesia
MeSH Terms: interventions — Phentolamine; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OraVerse (Experimental): OraVerse in doses of either 1/4, 1/2 or 1 cartridge (1.8mL)
  Interventions: Drug: OraVerse
- Sham injection (Sham Comparator): Dentist simulates injection with dental syringe
  Interventions: Other: Sham injection

INTERVENTIONS:
Drug: OraVerse — 1.8mL dental cartridge delivered in doses of either 1/4, 1/2 or 1 cartridge depending on subject weight
  Arms: OraVerse
Other: Sham injection — No drug administered, simulation of injection used in same manner as drug
  Arms: Sham injection

SUMMARY:
The purpose of this study is to determine whether OraVerse is safe and effective for the reversal of dental anesthesia in children 2 to 5 years of age weighing at least 10 kg.

DETAILED DESCRIPTION:
This Phase 4 clinical study is designed as a multicenter, randomized, double-blinded, controlled study to evaluate the safety and efficacy of OraVerse in approximately 150 children 2 to 5 years of age. OraVerse or sham injection is administered at the completion of a dental procedure requiring local anesthesia with lidocaine 2% with 1:100,000 epinephrine. The dental procedure(s) comprising restoration/fillings shall be performed in a single quadrant of the mouth.

The primary endpoint is safety and tolerability of OraVerse as measured by adverse events, vital signs, oral cavity assessments, nerve injury, and analgesics for intraoral pain. Secondary objectives in subjects 4 and 5 years of age include the safety and tolerability of OraVerse as measured by pain assessments using W-B PRS and evaluation of efficacy assessed by a pediatric Functional Assessment Battery (pFAB) and standardized lip and tongue palpation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 2 to 5 years of age
* Sufficiently healthy as determined by the Investigator to receive routine dental care
* Requires a restorative procedure (restoration/filling) in a single quadrant of the mouth
* Requires local anesthesia with lidocaine 2% with 1:100,000 epinephrine administered by submucosal injection
* For subjects undergoing mandibular procedures, require an inferior alveolar nerve block for the restorative procedure
* Dental procedure(s) completed within 60 minutes of injection of local anesthetic
* For subjects 4 and 5 years of age, can be trained in standardized lip/tongue palpation procedure and pFAB
* Subjects who are trainable in pFAB and standardized lip/tongue palpation procedure have either:

  * normal pFAB at baseline prior to administration of local anesthetic and
  * at least one abnormal function (smiling, speaking, drinking or drooling) at the completion of the dental procedure OR
  * normal lip sensation at baseline prior to administration of local anesthetic and
  * numbness of the relevant lip quadrant at completion of the dental procedure
* Subjects give written or verbal assent, as capable and appropriate, and parent(s) or legal guardian(s) give written informed consent

Exclusion Criteria:

* Weight less than 10 kg
* Weight less than 15 kg if 4 or 5 years of age
* History or presence of any condition that contraindicates routine dental care or use of local anesthetic
* Requires more than ¼ cartridge of local anesthetic if weight is ≥ 10 kg and < 15 kg, more than ½ cartridge of local anesthetic if weight is ≥ 15 kg and < 30 kg, and more than 1 cartridge of local anesthetic if weight is ≥ 30 kg, excluding supplemental injections
* Allergy or intolerance to lidocaine, epinephrine, sulfites, phentolamine, nitrous oxide or topical benzocaine
* Has used any investigational drug and/or participated in any clinical study within 30 days of study drug administration
* Has participated in this study or any previous study of phentolamine mesylate for reversal of local soft tissue anesthesia (STA)
* Any use of commercial OraVerse™ within 30 days of study drug administration
* Use of opioid or opioid-like analgesics within 24 hours prior to administration of local anesthetic
* Requires the use of local anesthetic other than lidocaine 2% with 1:100,000 epinephrine to perform the scheduled dental procedure
* Requires the use of general anesthesia or sedatives except for nitrous oxide to perform the scheduled dental procedure
* Any condition which in the opinion of the Investigator increases the risk to the subject of participating in this study or decreases the likelihood of compliance with the protocol

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2012-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Up to 3 days
Clinically significant changes in vital signs | Up to 3 days
  Blood pressure and pulse
Clinically significant changes in oral cavity assessments | Up to 3 days
Nerve injury | Up to 3 days
Analgesics required for intraoral pain | Up to 3 days

SECONDARY OUTCOMES:
incidence, severity and duration of intraoral pain as measured by W-B PRS | Up to 3 days
  Wong-Baker Pain Rating Scale used to assess subject pain
Time to normal function | Up to 3 days
  Measured by pediatric Functional Assessment Battery (pFAB) to determine when speaking, eating, drinking, drooling return to baseline
Time to normal lip sensation | Up to 3 days
  Measures time to normal lip and tongue sensation using standardized lip/tongue palpation procedure
Time to normal tongue sensation | Up to 3 days
  Measures time to normal tongue sensation using standardized lip/tongue palpation procedure

CONTACTS AND LOCATIONS:
Overall Officials: Paul Moore, DMD,PhD,MPH, Principal Investigator — University of Pittsburgh School of Dental Medicine; Elliot Hersh, DMD,MS,PhD, Principal Investigator — University of Pennsylvania; Joel Berg, DDS,MS, Principal Investigator — Seattle Children's Hospital; Judith Chin, DDS,MS, Principal Investigator — Indiana University; Brent Lin, DMD, Principal Investigator — University of California, San Francisco; Paul Casamassimo, MS,DDS, Principal Investigator — Nationwide Children's Hospital; Adam Marberger, DDS, Principal Investigator — Jean Brown Research
Locations (7):
- United States (7):
  - University of California, San Francisco, San Francisco, California
  - Indiana University School of Dentistry, Indianapolis, Indiana
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Pennsylvania School of Dental, Philadelphia, Pennsylvania
  - University of Pittsburgh School of Dental Medicine, Pittsburgh, Pennsylvania
  - Jean Brown Research, Salt Lake City, Utah
  - Center for Pediatric Dentistry, Seattle, Washington

REFERENCES:
- [Background] Hersh EV, Moore PA, Papas AS, Goodson JM, Navalta LA, Rogy S, Rutherford B, Yagiela JA; Soft Tissue Anesthesia Recovery Group. Reversal of soft-tissue local anesthesia with phentolamine mesylate in adolescents and adults. J Am Dent Assoc. 2008 Aug;139(8):1080-93. doi: 10.14219/jada.archive.2008.0311. PMID 18682623
- [Background] Moore PA, Hersh EV, Papas AS, Goodson JM, Yagiela JA, Rutherford B, Rogy S, Navalta L. Pharmacokinetics of lidocaine with epinephrine following local anesthesia reversal with phentolamine mesylate. Anesth Prog. 2008 Summer;55(2):40-8. doi: 10.2344/0003-3006(2008)55[40:POLWEF]2.0.CO;2. PMID 18547152
- [Background] Tavares M, Goodson JM, Studen-Pavlovich D, Yagiela JA, Navalta LA, Rogy S, Rutherford B, Gordon S, Papas AS; Soft Tissue Anesthesia Reversal Group. Reversal of soft-tissue local anesthesia with phentolamine mesylate in pediatric patients. J Am Dent Assoc. 2008 Aug;139(8):1095-104. doi: 10.14219/jada.archive.2008.0312. PMID 18682624
- [Background] Laviola M, McGavin SK, Freer GA, Plancich G, Woodbury SC, Marinkovich S, Morrison R, Reader A, Rutherford RB, Yagiela JA. Randomized study of phentolamine mesylate for reversal of local anesthesia. J Dent Res. 2008 Jul;87(7):635-9. doi: 10.1177/154405910808700717. PMID 18573982